CLINICAL TRIAL: NCT06411548
Title: Feasibility of a Bolus Calculator Without Carbohydrate Counting in Type 1 Diabetes Patients Under Multiple Daily Injections (MDI) Therapy: A Supervised Randomized Controlled Trial.
Brief Title: InsuLearn Feasibility With Type 1 Diabetes Patients Under MDI Therapy
Acronym: InsuLearn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Anas El Fathi, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 231610
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: InPen; Dexcom CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized crossover: Participants will be randomized to the order that they experience the use of InsuLearn (for 24 hours each, without washout in between): InsuLearn→UC or UC→InsuLearn. UC stands for usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- InsuLearn→Usual Care (Active Comparator): During the first 24 hours of the hotel admission (visit 6), participants' insulin dose will be calculated by the InsuLearn, MD approved, report. The second 24 hours of the hotel admission (visit 7), participants will use their usual care method to calculate their insulin dose.
  Interventions: Device: InsuLearn
- Usual Care→InsuLearn (Active Comparator): During the first 24 hours of the hotel admission (visit 6), participants' insulin dose will be calculated by their usual care method. The second 24 hours of the hotel admission (visit 7), participants will use the InsuLearn, MD approved, report to calculate their insulin dose.
  Interventions: Device: InsuLearn

INTERVENTIONS:
Device: InsuLearn — InsuLearn is an artificial intelligence (AI)-algorithm that analyses collected participants data: CGM, insulin, and meal categories to learn the optimal insulin dose. InsuLearn will run offline in a study laptop to generate the optimal insulin dose for each meal category. The algorithm will generate an ambulatory glucose profile (AGP) report with new settings for the InPen™ meal estimation bolus calculator. The study physician will review the report and the algorithm recommendations. The study physician can accept or modify the algorithm recommendations as per his judgment. The new settings will be used during the intervention admission.

SUMMARY:
This is a 24-hour, randomized, crossover, single-center trial where participants are randomized to either start with the InsuLearn intervention or the usual care (UC) intervention. In the InsuLearn intervention, insulin doses are optimized using data collected in a 4-weeks at home data collection period.

DETAILED DESCRIPTION:
Following recruitment and screening, 12 participants will be randomized to either the InsuLearn→UC or the UC→InsuLearn sequence. Participants will be trained in the use of a Continuous Glucose Monitor (CGM) (Dexcom G6 or Guardian™ 4), smart insulin pen (SIP, InPen™, Medtronic) and the InPen™ bolus calculator phone application. The InPen™ application will be set to the "meal estimation" mode where the user can select the meal category: if it is a breakfast/lunch/dinner/snack and if it has low/med/high carb amount. During the one-month data collection period, participants will be asked to use the InPen™ app to log and deliver their insulin doses. Before the hotel admission, InsuLearn will analyze the collected data to learn a new optimized insulin dose for each meal category. InsuLearn will generate a report of suggested new insulin doses that will be reviewed, approved, or changed by the study physician as needed. In the 24-h supervised interventions (hotel admission), the participant will consume three standardized meals, a med-carb lunch, a high-carb dinner, and low-carb breakfast. The insulin dose delivered in each admission will be either calculated by participants as per their UC or is as provided by the InsuLearn approved report. The two interventions are combined into a 2-day admission without a washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 years old at time of consent.
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year.
3. Hemoglobin A1c (HbA1c) between 6.5% - 10.0%, inclusive, within the past 60 days.
4. Currently using insulin under multiple daily injections (MDI) therapy for at least six months.
5. Willingness to wear the study continuous glucose monitor (CGM) during the duration of the study.
6. Access to the internet and willingness to upload data during the study as needed.
7. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
8. Investigator has confidence that the subject can successfully operate all study devices and can adhere to the protocol.
9. Willingness to remain on same dose of non-insulin glucose-lowering agent during the trial (including metformin/biguanides, GLP-1 receptor agonists, pramlintide, DPP-4 inhibitors, sulfonylureas and naturaceuticals).

Participant Exclusion Criteria

1. NPH (neutral protamine hagedorn) insulin
2. Use of any medication that at the discretion of the investigator is deemed to interfere with the trial.
3. Currently being treated for a seizure disorder.
4. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol, such as but not limited to, the following examples:

   1. Inpatient psychiatric treatment in the past 6 months
   2. Presence of a known adrenal disorder
   3. Abnormal liver function test results (Transaminase >3 times the upper limit of normal)
   4. Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2).
   5. Active gastroparesis requiring medical therapy.
   6. Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L).
   7. Abuse of alcohol or recreational drugs
   8. Infectious process not anticipated to be resolved prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis, deep tissue infection).
   9. Uncontrolled arterial hypertension (Resting diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg).
   10. Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy or VEGF inhibitor injections) in the past 12 months.
5. Currently pregnant or intent to become pregnant during the trial.
6. Currently breastfeeding.
7. An injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication, or disease in the judgment of the investigator will affect the completion of the protocol.
8. Participation in another pharmaceutical or device trial at the time of enrolment or during the study.
9. Non-stable dose of non-insulin glucose-lowering agent during the trial (including metformin/biguanides, GLP-1 receptor agonists, pramlintide, DPP-4 inhibitors, sulfonylureas and naturaceuticals) as defined by study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Low blood glucose index (LBGI) | Six hours after the three meals
  The primary outcome will be, per protocol (>70% of CGM values available after a meal), analysed using repeated measures ANOVA within-group contrast: i.e., InsuLearn vs. usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Anas Fathi, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the primary manuscript is published.
Access Criteria: The Data Sharing Agreements will be formulated by the study team